CLINICAL TRIAL: NCT02530554
Title: Pilot Trial Assessment of the Antimicrobial Efficacy of Medline 2% CHG Cloth Preoperative Skin Preparation
Brief Title: Pilot Trial of Chlorhexidine Gluconate (CHG) Preoperative Skin Preparation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R15-028
Record Dates: First submitted 2015-08-16; First posted 2015-08-21 (Estimated); Results first posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Surgery
Keywords: Preoperative surgical skin preparation
MeSH Terms: interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHG Cloth (Experimental): 3 min application time
  Interventions: Drug: CHG
- Comparator CHG (Active Comparator): Marketed 2% CHG
  Interventions: Drug: CHG

INTERVENTIONS:
Drug: CHG — Single application
  Other Names: Chlorhexidine Gluconate

SUMMARY:
Pilot study to evaluate and compare activity of CHG preoperative preparation with comparator CHG

DETAILED DESCRIPTION:
Evaluate and compare similar preoperative surgical preparations in healthy volunteers. Efficacy was assess using Tentative Final Monograph (TFM) criteria.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* No dermatological conditions

Exclusion Criteria:

* Sensitivity to CHG
* Sensitivity to natural latex rubber or adhesive skin products

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R Olsavszky, MD, Principal Investigator — S.C. Bio High Tech S.R.L

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Upon achieving sufficient microbial growth prior to product application on either the abdomen and groin regions, sites of the participant were then randomized to received two products for an evaluation or up to 4 sites.
Pre-assignment Details: Participants were randomized to be treated with at least 2 treatments/ Arms at the same time for both groin and abdomen. Total numbers represent participants.
Units Other Than Participants: Sites
Groups:
- CHG 3 Min Abdomen; CHG 3 Min Groin: 3 min application time
- Comparator CHG Abdomen: Comparator CHG on abdomen sites
- Comparator CHG Groin: Comparator CHG on groin sites
Period: Overall Study
Arm/Group | CHG 3 Min Abdomen | CHG 3 Min Groin | Comparator CHG Abdomen | Comparator CHG Groin
Started (14 total participants,12 treated on all 4 sites & 2 treated on 2 sites with both interventions.) | 12; 12 Sites | 14; 14 Sites | 12; 12 Sites | 14; 14 Sites
Completed | 12; 12 Sites | 14; 14 Sites | 12; 12 Sites | 14; 14 Sites
Not Completed | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites | 0; 0 Sites

BASELINE CHARACTERISTICS:
Population: Participants would receive up to 2 different treatments at the same time. Treatments included CHG 3 min or comparator CHG.
Groups:
- CHG 3 Min, Comparator CHG: CHG applied for 3 min, Comparator CHG applied per instructions.
Arm/Group | CHG 3 Min, Comparator CHG
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 56 [24 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 3
Region of Enrollment [Number; unit: participants]
  Romania | 14

OUTCOME MEASURES:

1. Primary Outcome: Log Change in Bacterial Flora on Abdomen and Groin
Description: Change was calculated as the baseline time point minus the later time points over an 8 hour period.
Time Frame: 10 min, 6 hr and 8 hr
Measure: Mean (95% Confidence Interval); unit: Log (CFU)
Units Other Than Participants: Sites
Groups:
- Comparator CHG Abdomen: CHG comparator applied to abdomen
- Comparator CHG Groin: CHG Comparator applied to groin
Arm/Group | CHG 3 Min Abdomen | CHG 3 Min Groin | Comparator CHG Abdomen | Comparator CHG Groin
Number analyzed (Participants) | 12 | 14 | 12 | 14
Number analyzed (Sites) | 12 | 14 | 14 | 14
Log (CFU)
  10 min | 2.9 [2.1 to 3.7] | 3.7 [3.0 to 4.4] | 2.3 [1.5 to 3.1] | 3.0 [2.3 to 3.7]
  6 hour | 2.9 [2.1 to 3.6] | 3.9 [3.2 to 4.7] | 2.5 [1.7 to 3.3] | 3.3 [2.6 to 4.1]
  8 hour | 2.9 [2.2 to 3.6] | 4.6 [3.9 to 5.3] | 2.3 [1.5 to 3.0] | 3.3 [2.7 to 4.0]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from baseline out to 8 hours.
Description: Participants received up to 2 products at the same time.
Groups:
- CHG 3 Min and Comparator CHG: 3 min application time for CHG and the comparator CHG was applied according to instructions.
Arm/Group | CHG 3 Min and Comparator CHG
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidential information as part of the contract.